CLINICAL TRIAL: NCT03107767
Title: The PRO-malleol Study
Brief Title: Study of Re-operation Rate After Introduction of Evidence Based Algorithm for the Treatment of Ankle Fractures
Acronym: PRO-Malleol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Peter Toft Tengberg, Consultant, PhD, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO-Malleol study
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Ankle Fractures; Surgery; Syndesmotic Injuries; Posterior Malleolus Fractures
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries

STUDY DESIGN:
Intervention Model Description: A prospective cohort, following the introduction of an evidence based algorithm, will be compared to a matched historical cohort from the previous years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Cohort (Active Comparator): The prospective cohort following introduction of the evidence based algorithm for ankle fractures.
  Interventions: Procedure: PRO-malleol algorithm
- Historical Cohort (No Intervention): Patients treated before introduction of algorithm. Matched to prospective cohort for comparison

INTERVENTIONS:
Procedure: PRO-malleol algorithm — An evidence based algorithm for ankle fractures
  Arms: Prospective Cohort

SUMMARY:
There is a high incidence of re-operations after surgery for ankle fractures. According to the Danish Fracture Database (DFDB) the re-operation rate, excluding hardware removal, is almost 10%.

We are conducting a study on the efficacy of an evidence based algorithm for the treatment of ankle fractures.

DETAILED DESCRIPTION:
Treatment of ankle fractures is complex and includes assessment of fracture pattern, severity of soft-tissue involvement and general health- and functional status of the patients. Historically most fractures, undisplaced as well as displaced, were treated non-operatively with acceptable results but in recent years there is an increasing trend towards operative management of unstable fractures. Techniques for operative management of ankle fractures are varied and assessment of instability is mainly based on classic x-ray classification systems such as Lauge-Hansen or the AO that are difficult to reproduce[6].

We hypothesize that a standardized and evidence based approach to ankle fracture management will lead to a decrease in re-operation rate.

The aim of this study is to standardize the management of ankle fractures in our department, by introducing an algorithm based on best evidence present. We want to investigate:

1. The effect of this algorithm on the re-operation rate of surgically treated ankle fractures in a two-year prospective observational setup with a minimum of one-year of follow-up.
2. The need for surgery and functional outcome of patients with isolated lateral malleolus fractures in which the treatment is dictated by ankle stability assessed on weight bearing radiographs.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated for ankle fractures at our institution during the study period are asked to participate in the study.

Exclusion Criteria:

* Not speaking danish Not followed up at our institution Not mentally capable of filling out questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in re-operation rate | one year
  Change in re-operation rate following introduction of PRO malleol algorithm
Rate of surgery for isolated lateral ankle fractures | one year
  Rate of surgery for isolated lateral ankle fractures, following introduction of algorithm

SECONDARY OUTCOMES:
SF 36 | day 0 and 12 months
  SF 36 before fracture and at 12 months
Ollerud Molander Ankle Score | Before fracture, 6 weeks, 12 weeks and 1 year
Forgotten Joint Score | Before fracture, 6 weeks, 12 weeks and 1 year
  Before fracture, 6 weeks, 12 weeks and 1 year
Rate of complications not requiring surgery | One year
  DVT, Nerve damage,

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data will be anonymized and openly shared with any who requests it, after study publication.